CLINICAL TRIAL: NCT03002883
Title: Sacramento Taking Action Against Nicotine Dependence (STAND) at Sacramento City College
Brief Title: STAND Community College Tobacco Cessation Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Tobacco Related Disease Research Program (Other); Breathe California of Sacramento-Emigrant Trails (Unknown); Sacramento City College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 491744; 22BT-0057 (Other: Other)
Record Dates: First submitted 2016-12-19; First posted 2016-12-26 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (Placebo Comparator): Students referred to student health for tobacco cessation resources including campus "Quit Kits"
  Interventions: Behavioral: Usual Care
- Brief Motivational Interviewing (Active Comparator): Students received brief motivational interviewing by a student peer educator about tobacco cessation
  Interventions: Behavioral: Usual Care; Behavioral: Brief Motivational Interviewing
- Direct referral to quitline (Active Comparator): Students were directly referred to the state quitline for follow-up counseling
  Interventions: Behavioral: Usual Care; Behavioral: Direct referral to quitline

INTERVENTIONS:
Behavioral: Usual Care — Participant provided "Quit Kit" water bottle with small cessation aids (eg. sunflower seeds) and educated about student health as a cessation resource
Behavioral: Brief Motivational Interviewing — Peer educator conducts brief motivational interviewing about smoking cessation and participant goals
  Arms: Brief Motivational Interviewing
Behavioral: Direct referral to quitline — Peer educator educates about state quitline services and gets verbal consent to use quitline's direct referral web portal for quitline to contact participant in 1-2 business days about free counseling services to make a quit plan
  Arms: Direct referral to quitline

SUMMARY:
Community colleges have 45% of the nation's undergraduates and have a higher smoking prevalence rate than 4-year colleges. California's community colleges comprise the nation's largest higher education system, and Sacramento has the second largest community college district. As more colleges are encouraged to become smoke and tobacco-free campuses, smokers enrolled at community college campuses need greater support. However, community colleges may lack the student health clinic resources that 4-year colleges have for students who live on campus. Little evidence to date demonstrates effective interventions for smokers on community college campuses.

This pilot study seeks to demonstrate the feasibility and promising outcomes of two cessation interventions, compared with usual care on a community college campus. The first intervention was based on a promising model of brief motivational interviewing delivered by peer educators, developed by the community lead Breathe California of Sacramento-Emigrant Trails (BCSET) through the Sacramento Taking Action Against Tobacco Dependence (STAND) project. The second intervention was based on direct enrollment into the California Smokers' Helpline, which has demonstrated utility for promoting smoking cessation among young adults with low socioeconomic status. Usual care consisted of students going to the student health center for smoking cessation assistance.

ELIGIBILITY:
Inclusion Criteria:

* adult 18 years or older
* current smoker in the past 30 days
* smoker wants to quit
* smoker not currently participating in other smoking cessation activities, and
* smoker must be willing to accept randomization into any of the 3 study arms

Exclusion Criteria:

* students not proficient in communicating in English
* adults unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Biochemically validated smoking cessation | 6 months
  Point prevalence abstinence validated by saliva cotinine level

SECONDARY OUTCOMES:
Self-reported smoking cessation | 6 months
  Point prevalence abstinence by self-report on survey
Self-reported smoking cessation | 3 months
  Point prevalence abstinence by self-report on survey
Self-reported smoking cessation | 1 month
  Point prevalence abstinence by self-report on survey

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Tong, MD, Principal Investigator — University of California, Davis

IPD SHARING:
Plan to Share IPD: No